CLINICAL TRIAL: NCT04804969
Title: MyoVista wavECG Clinical Validation Study
Brief Title: MyoVista wavECG Clinical Validation Study Versus Low e' on Echocardiogram
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Heart Test Laboratories, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HS-CLINVAL-001
Record Dates: First submitted 2021-03-16; First posted 2021-03-18 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Cardiac Disease
Keywords: Left Ventricular Diastolic Dysfunction; Electrocardiograph
MeSH Terms: conditions — Heart Diseases; Ventricular Dysfunction, Left

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- At Risk Echo Referrals: Study subjects will be drawn from patients who are at-risk for cardiac disease and who have been referred for 2D transthoracic echocardiogram as standard of care. All will receive a MyoVista wavECG test.
  Interventions: Device: MyoVista wavECG Test

INTERVENTIONS:
Device: MyoVista wavECG Test — The MyoVista wavECG is a standard 12-Lead high-performance, multi-channel resting interpretive electrocardiograph providing both a Glasgow Interpretive Analysis and unique MyoVista wavECG Information.

SUMMARY:
Clinical validation study of the MyoVista wavECG.

DETAILED DESCRIPTION:
This is a multi-center, non-interventional, single arm clinical study of the MyoVista wavECG for the detection of LV relaxation abnormalities. Study subjects will be drawn from patients who are at-risk for cardiac disease and who have been referred for 2D transthoracic echocardiogram.

The study will be conducted at a minimum of three investigational sites within the United States.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with risk factors for cardiac disease or suspected of having cardiac disease during clinical assessment.
* The subject provides written informed consent using an Informed Consent Form that is reviewed and approved by the site's Institutional Review Board (IRB).
* Conventional ECG results show a sinus rhythm and no other contraindicated rhythm abnormalities (see exclusions below).
* Subject is >/= 22 years of age

Exclusion Criteria:

* The subject has current acute coronary syndrome, decompensated heart failure or stroke
* The subject has received any prior cardiac interventions or surgical therapeutic procedures relating to cardiac abnormalities: valve replacement, pacemaker implantation, coronary artery bypass grafting (CABG), heart transplant, ablation, coronary stent placement, etc.
* Conventional ECG results indicating a lack of sinus rhythm and/or any other contraindicated rhythm abnormalities, including: active atrial fibrillation or atrial flutter, left anterior fascicular block, left and/or right bundle branch block
* The subject is pregnant at the time of the study testing
* The subject has chest deformities that interfere with accurate measurement of ECG (either conventional or wavECG)
* Subjects with central nervous system or musculoskeletal abnormalities that may interfere with accurate acquisition of ECG and/or echocardiogram measurements.
* The subject is enrolled in another clinical study that may interfere with MyoVista or echocardiogram measurements. Exceptions to this may be approved by HeartSciences.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with risk factors for cardiac disease or suspected of having cardiac disease during clinical assessment and have been referred to the site for 2D transthoracic echocardiogram.
Sampling Method: Non-Probability Sample
Enrollment: 575 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity | Baseline
  Sensitivity and specificity of the MyoVista for the classification of Low e' from echocardiogram where a "positive" includes Positive and Highly Positive MyoVista Device outcomes.

SECONDARY OUTCOMES:
Sensitivity and Specificity | Baseline
  Sensitivity and specificity of the MyoVista for classification of Low e' versus echocardiogram where a "positive" includes Borderline, Positive and Highly Positive MyoVista Device outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Partho Sengupta, MD, Principal Investigator — Robert Wood Johnson University Hospital
Locations (5):
- United States (5):
  - Scripps Memorial Hospital, La Jolla, California
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Montefiore Medical Center, The Bronx, New York
  - Einstein Medical Center, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No